CLINICAL TRIAL: NCT04727242
Title: Phase 2 Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) With Gemcitabine Followed by Systemic Adjuvant Chemotherapy With Dacarbazine for Locally Recurrent Uterine Leiomyosarcoma (LMS)
Brief Title: CytoreductiveSurgery & HIPEC w/Gemcitabine+Chemotherapy w/Dacarbazine in Uterine Leiomyosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-56728; SARCOMA0045 (Other: OnCore); NCI-2021-03258 (Other: CTRP)
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: LMS - Leiomyosarcoma; Uterine Leiomyosarcoma
MeSH Terms: interventions — Gemcitabine; Dacarbazine; Cytoreduction Surgical Procedures; Magnetic Resonance Spectroscopy; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cytoreductive Surgery+HIPEC gemcitabine+dacarbazine (Experimental): * Cytoreductive surgery followed by hyperthermic intraperitoneal chemotherapy (HIPEC) with gemcitabine followed by postoperative systemic chemotherapy with dacarbazine. Conceptually, HIPEC will be administered as a 60 minute heated intraperitoneal infusion (ie, intraperitoneal "wash" or "lavage").
  * HIPEC: Gemcitabine will be instilled at a dose of 1000 mg/m2 for 60 minutes at temperatures of 42° to 43°C.
  * Systemic adjuvant chemotherapy starting 30 days ± 14 days post surgery. Dacarbazine 1000 mg/m2 IV every 3 weeks x 6 cycles
  Interventions: Drug: Gemcitabine; Drug: Dacarbazine; Procedure: Cytoreductive Surgery; Behavioral: Functional Assessment of Cancer Therapy (FACT) G questionnaire; Procedure: Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) Scan; Drug: Gadolinium

INTERVENTIONS:
Drug: Gemcitabine — Hyperthermic intraperitoneal chemotherapy (HIPEC) with gemcitabine. Gemcitabine will be instilled at a dose of 1000 mg/m2 for 60 minutes at temperatures of 42° to 43°C.
  Other Names: Gemzar; Infugem; difluorodeoxycytidine hydrochloride
Drug: Dacarbazine — Dacarbazine 1000 mg/m2 IV every 3 weeks x 6 cycles given IV
  Other Names: Dimethyl (triazeno) imidazolecarboxamide; Dacarbazine - DTIC; Biocarbazine
Procedure: Cytoreductive Surgery — Surgery for cancer removal
Behavioral: Functional Assessment of Cancer Therapy (FACT) G questionnaire — Preoperative and Postoperative FACT G questionnaire to assess QoL
Procedure: Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) Scan — Radiologic imaging after Cycle 3 and 6 and at each follow up visit
Drug: Gadolinium — Contrast Agent

SUMMARY:
The purpose of this study is to find out if giving a dose of heated chemotherapy in the abdomen immediately after surgery that is done to remove uterine leiomyosarcoma type of cancer will help lower the risk of the cancer coming back in the future.

DETAILED DESCRIPTION:
Primary Objective:

- To assess the efficacy of cytoreductive surgery with gemcitabine HIPEC followed by postoperative systemic chemotherapy with dacarbazine in subjects with locally recurrent uterine LMS.

Secondary Objectives:

* To assess the safety of cytoreductive surgery with gemcitabine HIPEC in subjects with locally recurrent uterine LMS.
* To assess the 6 month and 12 month intraabdominal relapse free survival in subjects with locally recurrent uterine LMS
* To determine quality of life prior to therapy (within 28 days prior to surgery with HIPEC), 4 to 6 weeks after surgery with HIPEC, and then at Cycle

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of uterine leiomyosarcoma (LMS) with evidence of local recurrence.
2. Imaging provides evidence of locally recurrent uterine LMS.
3. Candidate for potentially radical, maximal effort cytoreductive surgery at the discretion and expertise of the treating physician.
4. Age ≥ 18 years.
5. Life expectancy > 3 months.
6. Women of childbearing potential (WOCBP) will have a negative pregnancy test ≤ 7 days prior to surgery (this test can be omitted if subject is post menopausal by either surgery or elevated FSH)
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
8. Hemoglobin (HGB) ≥ 9 g/dL.
9. White blood cell count (WBC) ≥ 3.0 K/ul.
10. Absolute neutrophil count (ANC) ≥ 1.5 K/ul.
11. Platelets (PLT) ≥ 100 K/ul.
12. Total bilirubin within normal institutional limits.
13. Serum glutamic oxaloacetic transaminase (SGOT/Serum glutamic pyruvic transaminase (SGPT) < 2.5 x institutional upper limit of normal (ULN).
14. Creatinine < 1.5 x ULN or creatinine clearance > 60 mL/min according to Cockroft Gault formula.
15. Prothrombin Time (PT) such that international normalized ratio (INR) is < 1.5 (or an in range INR, usually between 2 and 3, if a subject is on a stable dose of therapeutic warfarin or low molecular weight heparin) and a partial thromboplastin time (PTT) < 1.2 times control.
16. Serum albumin ≥ 2.5 g/dL.
17. Ability to understand and the willingness to personally sign the written IRB approved informed consent document.

Note that this study does not allow the use of a legally authorized representative

Exclusion Criteria:

1. Recurrence of LMS within less than 6 months after the last dose of gemcitabine.
2. Active extra abdominal disease including active malignant pleural effusion. Subjects who have been successfully treated with neoadjuvant chemotherapy and no longer have (malignant) pleural effusions may be included.
3. Prior gemcitabine given in non adjuvant setting.
4. Prior treatment with dacarbazine.
5. Active infection requiring antibiotics.
6. Unresolved toxic effects of prior therapy (except alopecia). Resolution is considered ≤ Grade 1 per NCI CTCAE, version 5.0.
7. Pregnant.
8. Breast feeding.
9. Presence of metastatic liver disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 1 year
  Progression free survival as measured from the time of surgery until death or disease progression.

SECONDARY OUTCOMES:
Rate of Grade 4 infections | 30 days post surgery with gemcitabine HIPEC
  Rate of Grade 4 infections within 30 days post surgery with gemcitabine HIPEC will be assessed using CTCAE version 5.0.
Intraabdominal relapse free survival | 6 months
  Relapse free survival as measured from time of surgery until intraabdominal recurrence
Intraabdominal relapse free survival | 12 months
  Relapse free survival as measured from time of surgery until intraabdominal recurrence
Overall Functional Assessment of Cancer Therapy: General (FACT G) score | Baseline, 4 to 6 weeks post-surgery with HIPEC
  Difference in overall FACT G score from baseline to 4 to 6 weeks post-surgery with gemcitabine HIPEC.
  FACT G is a quality of life questionnaire composed of 27 items divided into four main quality of life categories: Physical Well Being (PWB); Social/Family Well Being (SWB); Emotional Well Being (EWB); and Functional Well Being (FWB). Total FACT G score is obtained by summing the scores from the four main QoL categories (PWB; SWB; EWB; FWB). The range of the scale is 0-108. Negatively worded items are reverse scored prior to summing so that higher subscale and total scores indicate better Quality of life (Qol).

CONTACTS AND LOCATIONS:
Overall Officials: Kristen N Ganjoo, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No